CLINICAL TRIAL: NCT04625192
Title: Lateral Sinus Lift Technique Using Trephine Osteotomy With Simultaneous Implant Placement (Clinical Trial)
Brief Title: Trephine Osteotomy in Lateral Sinus Lift
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Trephine osteotomy
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Sinus Lift

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sinus lifting with trephine osteotomy (Experimental)
  Interventions: Procedure: Trephine osteotomy

INTERVENTIONS:
Procedure: Trephine osteotomy — * Using a trephine on a straight implant handpiece (at approximately 1800 rpm) with copious irrigation to avoid overheating the bone, a round bone cut will be made 4 -5 mm above the crest of the alveolar ridge.
  * The trephine is positioned perpendicular to the lateral wall, removing the outer cortex with a very gentle touch to avoid tearing the schneiderian membrane.

SUMMARY:
Trephine osteotomy was used for lateral sinus lifting technique associated with sinus floor augmentation using the autogenous bone resulting from implant drilling using specialized trephine drills.

DETAILED DESCRIPTION:
The study includes 14 patients in whom the lateral sinus lift technique was performed using the trephine osteotomy with simultaneous implant placement.

Sinus floor augmentation with autogenous bone graft resulting from implant site preparation with trephine drills.

Implant stability and rate of complications such as Schneiderian membrane perforation and bleeding will be assessed.

Patients will also provide their subjective assessment of postoperative pain and swelling. Vertical bone height, that will be gained, will be assessed radiographically

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders requiring implant placement in the posterior maxilla.
* Age between 20-50 years.
* Tooth extractions at the implant sites were performed at least 4 months before surgery.
* Residual bone height between the alveolar bone crest and the sinus floor ranges from 4 to 6 mm.
* Patients who are willing and fully capable to comply with the study protocol

Exclusion Criteria:

* Maxillary sinus pathologies (sinusitis, long standing nasal obstruction)
* Any disease contraindicating surgery (e.g. uncontrolled diabetes)
* Heavy smokers
* Acute oral infections
* Poor oral hygiene
* A history of radiotherapy or chemotherapy of the head and neck region

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in Implant stability | at baseline and 6 months
  This will be measured by implant stability meter (OsstellTM)
change in bone density | at baseline, 3rd and 6th months
  Panoramic radiography will be performed immediately postoperatively and cone beam computed tomography (CBCT)
change in bone volume | at baseline, 3rd and 6th months
  Panoramic radiography will be performed immediately postoperatively and cone beam computed tomography (CBCT)
change in bone vertical bone height | at baseline, 3rd and 6th months
  Panoramic radiography will be performed immediately postoperatively and cone beam computed tomography (CBCT)

SECONDARY OUTCOMES:
post operative pain | after 1 week
  This will be assessed using a 10-point Visual Analogue Scale (VAS) in the 1st week postoperatively.
  (0-1=None, 2-4=Mild-Moderate, 8-10= Severe)
Postoperative edema | after 1 week
  * None (no inflammation).
  * Mild (intraoral swelling confined to the surgical field).
  * Moderate (extraoral swelling in the surgical zone).
  * Severe (extraoral swelling spreading beyond the surgical zone

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt